CLINICAL TRIAL: NCT07278102
Title: A Korean Multicenter Prospective Observational Study on Efficacy of 90Y for Hepatocellular Carcinoma-early Stage
Brief Title: A Prospective Observational Study on Efficacy of TARE for Early Stage HCC
Acronym: KURE-YTT-HCC
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government); Severance Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yoon Jun Kim, Professor, Seoul National University Hospital
Other Study IDs: KURE-YTT-HCC
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Radioembolization; Hepatocellular Carcinoma (HCC); Early Stage
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TARE: early stage hepatocellular carcinoma
  Interventions: Procedure: transarterial radioembolization

INTERVENTIONS:
Procedure: transarterial radioembolization — TARE with 90Y

SUMMARY:
The aim of the current study is to analyze treatment outcomes (best target lesion response, overall survival, time to target lesion progression, time to overall progression, and treatment-related adverse event) using prospectively collected clinical and imaging data in patients with BCLC 0 or A HCCs treated with TheraSphere® in four large-volume hospitals from Korea. The results will pave the way for expanding 90Y-TARE indication and refining reimbursement guidelines, and provide baseline data for possible subsequent future studies.

ELIGIBILITY:
Inclusion Criteria:

* A. Patients receiving TARE using TheraSphere® B. Treatment naïve BCLC 0 or A single HCC up to 8 cm (diagnosed according to diagnostic criteria of KLCA-NCC) C. Tumor involvement < 50% of total liver volume based on dynamic CT or MRI D. Age > or = 18 E. ECOG performance status 0 F. AST/ALT < or = 5 times the upper limits of normal G. A life expectancy > 3 months H. Non-pregnant with an acceptable contraception in premenopausal women I. Ability to provide written informed consent and to comply with all study conditions

Exclusion Criteria:

* A. Contraindications to angiography and selective catheterization B. Known anaphylaxis to iodinated contrast C. Expected lung dose > 30Gy per a session D. Unable to avoid non-target 90Y flow into the extrahepatic organs except the lungs E. Decompensated liver cirrhosis (Child-Pugh score > 7) F. Active uncontrolled infection G. Pregnancy H. Current or history (< or = 5 years) of malignancies in the other organs I. History of liver transplantation J. Any vascular invasion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving TARE using TheraSphere® Treatment naïve BCLC 0 or A single HCC up to 8 cm (diagnosed according to diagnostic criteria of KLCA-NCC) Tumor involvement < 50% of total liver volume based on dynamic CT or MRI Age > or = 18 ECOG performance status 0 AST/ALT < or = 5 times the upper limits of normal A life expectancy > 3 months Non-pregnant with an acceptable contraception in premenopausal women Ability to provide written informed consent and to comply with all study conditions
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From enrollment to the end of treatment at 3 years
  Overall survival
best target lesion response | "From enrollment to the end of treatment at 3 years
  best target lesion response

SECONDARY OUTCOMES:
Time to target lesion progression | From enrollment to the end of treatment at 3 years
  Time to target lesion progression
Time to overall progression | From enrollment to the end of treatment at 3 years
  Time to overall progression
Treatment-related adverse events rates | From enrollment to the end of treatment at 3 years
  Treatment-related adverse events rates

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.tarekorea.com/company/02/